CLINICAL TRIAL: NCT05740631
Title: The Effect of Obeticholic Acid on Gut Microbiota, Gastric Motility, Accommodation, Gastrointestinal Peptide in Healthy Volunteers
Brief Title: The Effect of Obeticholic Acid in Healthy Volunteers
Acronym: OCARINA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Intercept Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Prof Dr Jan Tack, Head Division of Gastroenterology and Hepatology, Leuven University, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: S64643; 2020-004180-13 (EudraCT Number)
Record Dates: First submitted 2022-09-16; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Healthy
Keywords: Obeticholic acid; Farnesoid X receptor; gastric accommodation; gastrointestinal hormones; gut microbiota
MeSH Terms: interventions — obeticholic acid; Starch

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obeticholic acid (Experimental): FXR agonist, orally administration (10 mg)
  Assignment of treatment (placebo and obeticholic acid) will be randomized before study visit 1. Either placebo or obeticholic acid will be administered orally in a single-blind fashion for 21 days. After a washout period of 28 days, either placebo or obeticholic acid will be administered as appropriate for an additional 21 days.
  Interventions: Drug: Ocaliva
- Placebo (Placebo Comparator): Assignment of treatment (placebo and obeticholic acid) will be randomized before study visit 1. Either placebo or obeticholic acid will be administered orally in a single-blind fashion for 21 days. After a washout period of 28 days, either placebo or obeticholic acid will be administered as appropriate for an additional 21 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ocaliva — Assignment of treatment obeticholic acid will be started (randomized) after the study visit and administered orally in a single-blind fashion for 21 days.
  Other Names: obeticholic acid
  Arms: Obeticholic acid
Drug: Placebo — Assignment of treatment placebo will be started (randomized) after the study visit and placebo will be administered orally in a single-blind fashion for 21 days.
  Other Names: Placebo Oral Tablet (Starch)
  Arms: Placebo

SUMMARY:
This study investigates whether obeticholic acid affects gut microbiota, gastric motility, accommodation, and gastrointestinal peptide in healthy subjects.

This study is a single-blind, placebo-controlled, randomized study. Twelve healthy volunteers will take one tablet containing obeticholic acid (10 mg) or a placebo once per day for 21 days for the first intervention. After 28 days washout period, they will take a tablet different from the one taken in the first intervention.

Before the first intervention, they will receive MMC, IGP and endoscopy exam. At the end of the first and second interventions, they will receive the same exams. During MMC&IGP, we will take blood samples to measure plasma hormones (motilin, octa-ghrelin, GLP-1, GLP-2, GIP, and insulin) and take duodenal fluid. When the endoscopy, we will take samples from the duodenal for microbiota, permeability measurement, RNA, protein, and pathology.

Before and during the interventions, stool samples will be collected.

DETAILED DESCRIPTION:
Functional dyspepsia (FD) is a common functional gastroduodenal disorder that has a great social and economic impact on patients. The pathophysiology of FD remains poorly understood and is most likely heterogeneous, but likely candidates are genetic factors, stress and duodenal luminal factors, including bile acids. Obeticholic acid (OCA), a Farnesoid X receptor (FXR) agonist, is an effective drug for primary biliary cirrhosis. Recently, it has been shown that OCA altered the gut microbiome via induction of lower endogenous bile acid levels in mice. OCA might alter the gut microbiota and duodenal inflammation. Moreover, gastric motility, accommodation and gastrointestinal peptide might be affected through the change in duodenal circumstances. Therefore, the aim of the current research protocol is to investigate the relationship between FXR agonist and gut microbiota, gastric motility, accommodation, and gastrointestinal peptide in healthy volunteers. During the screening of our healthy volunteers, the study will be explained, and the informed consent will be read together. When the volunteer agrees, it will be checked whether the volunteer is included, and some questionnaires will also be completed. A total of 20 healthy volunteers will be included and then randomized. All volunteers participate in both treatment arms: OCA or placebo. Participants will take each OCA and placebo for 21 days across the washout period at home. A motility test is performed before and at the end of each treatment. A high-resolution pressure gauge (HRM) catheter is placed into the proximal part of the small intestine (checked by fluoroscopy) and an intravenous catheter in the arm for blood sampling. The measurement in the fasted state will be performed until a characteristic cycle called as migrating motor complex cycle (MMC) is measured at least once. During migrating motor complex measurement, blood samples will be taken via a syringe that we connect to the line of your catheter every 20 min within the first 60min of MMC measurement, then every 10 min until the end of MMC phase III. Duodenal fluids are also aspirated and collected during the fasted state. From 30 minutes after the end of the MMC measurement, participants will start to drink a liquid nutrient meal at a constant speed while gastrointestinal motility continues to be monitored. In the meantime, a blood sample is taken every 10 minutes to measure hormones later. The measurement will finish 60 minutes after the start of the meal. During intragastric pressure measurement, participants must score their appetite feelings every 5 minutes on a scale questionnaire. An endoscopy is performed before and at the end of each treatment. Duodenal tissues (maximum 9) are collected using biopsy forceps via an endoscope. Participants will collect stool samples at home using the sampling material before taking the drug on day 1 and after taking the drug on days 2, 4, 7, 14, and 21.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
2. Use of highly effective methods of birth control; defined as those that, alone or in combination, result in low failure rate (i.e., less than 1% per year) when used consistently and correctly; such as implants, injectables, combined oral contraceptives, some IUDs, true sexual abstinence (i.e. refraining from heterosexual intercourse during the entire period of risk associated with the Trial treatment(s)) or commitment to a vasectomised partner.
3. Subject is between 18 and 65 years of age
4. Subject has a BMI between 18 and 25 kg/m²

Exclusion Criteria:

1. Participant has a history of gastrointestinal or other significant somatic or psychiatric diseases or drug allergies, diabetes, a significant heart, lung, liver or kidney disease, a neurological disorder, abdominal surgery (including gallbladder removal, but those having undergone a simple appendectomy more than 1 year prior to the screening visit may participate),
2. Any disorder, which in the Investigator's opinion might jeopardise the participant's safety or compliance with the protocol
3. Any prior or concomitant treatment(s) that might jeopardise the participant's safety or that would compromise the integrity of the Trial
4. Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate, highly effective contraceptive
5. Participation in an interventional Trial with an investigational medicinal product (IMP) or device
6. High caffeine intake (> 500 ml coffee daily or equivalent).
7. Subject consumes excessive amounts of alcohol, defined as >21 units per week for men, >14 units per week for women.
8. Subject is currently (defined as within approximately 1 year of the screening visit) a regular or irregular user (including "recreational use") of any illicit drugs (including marijuana) or has a history of drug (including alcohol) abuse. Further, patient is unwilling to refrain from the use of drugs during this study.
9. Inability or unwillingness to perform all of the study procedures, or the subject is considered unsuitable in any way by the principal investigator.
10. Recent participation (<30 days) or simultaneous participation in another clinical study.
11. Prior participation in a clinical trial of obeticholic acid

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-07-22 (Estimated); Study Completion 2023-07-22 (Estimated)

PRIMARY OUTCOMES:
Changes in appetite after administration of obeticholic acid compared to placebo | During MMCⅢ (300 min)
  Assessment by questionnaire(100mm Visual Analogue Scale) every 10 minutes.

SECONDARY OUTCOMES:
Change in serum GI hormones concentrations | During MMCⅢ (300 min)
  Blood samples to assess GI hormones concentrations
Change in gastric motility | During MMCⅢ (300 min)
  IGP(Intragastric pressure) will be measured.
Change in gut microbiota | 12 days
  Stool samples will be collected for analyze gut microbiota.

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT05740631/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/31/NCT05740631/ICF_001.pdf